CLINICAL TRIAL: NCT02547389
Title: Enhancing Medical Compliance and Health-related Quality of Life of Patients With Epilepsy: Randomized Controlled Trial
Brief Title: Enhancing Medical Compliance and Health-related Quality of Life of Patients With Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Macmillan Research Group UK (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: nmp/22181
Record Dates: First submitted 2015-09-02; First posted 2015-09-11 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (IG) (Active Comparator): IG additionally received community health programs with health workers(intensive education, consultation services, maintenance of anepilepsy tracking card, and repeated reminders).
  Interventions: Behavioral: Community support group
- Control Group (CG) (Other): Patients in the CG were supplied with only printed epilepsy educational module
  Interventions: Other: Printed material Supported

INTERVENTIONS:
Behavioral: Community support group
  Arms: Intervention Group (IG)
Other: Printed material Supported
  Arms: Control Group (CG)

SUMMARY:
Improving medical compliance and health-related quality of life (HRQoL) among people with epilepsy (PWE) has become the focus of various treatment programs and behavioral interventions which continue to be challenging to both patients and health care professionals.

In order to design an effective intervention on the management of epilepsy, the drug management of epilepsy by community health workers was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants must have a definitive diagnosis of epilepsy for at least 6 months, based on the clinical judgement of the investigators. Epilepsy is defined by two or more unprovoked seizures. Clinical history, electroencephalography, and imaging data are all instrumental in rendering a formal decision. The seizure type, frequency, or severity are not criteria for exclusion, although this information will be recorded.
* Patients must have a seizure frequency of at least two seizures in a 6 month period of time.
* Patients must be on at least one anti-epileptic medication.
* Patients must be able to report seizure frequency with either a paper or electronic diary.
* Patients must be able to read and understand either English or Hindi.
* Patients must be able to complete questionnaires and provide informed consent to this study.

Exclusion Criteria:

* A diagnosis of psychogenic nonepileptic seizures
* Severe depression, anxiety, or psychosis
* Recent problem with substance abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Compliance with taking prescribed medications | 12 months
  Assessment of compliance with taking medications at regularly scheduled intervals

SECONDARY OUTCOMES:
Seizure frequency per month | change from baseline to 12 months in number of seizures per month assessed by patients diary
  Assessment of seizure count accuracy by assessing total number of seizures reported per month
Quality of Life (Malay Quality of Life in Epilepsy Inventory-30) | change from baseline to 12 months in quality of life assessed by Malay Quality of Life in Epilepsy Inventory-30
  Malay Quality of Life in Epilepsy Inventory-30, to assess for overall change in quality of life measures

CONTACTS AND LOCATIONS:
Overall Officials: Hitesh K Nayak, Principal Investigator — NMP Medical Research Institute; Neha Sharma, PhD, Study Director — Macmillan Research Group UK